CLINICAL TRIAL: NCT04353895
Title: Fluoro-registered Mazor X Stealth Edition Versus O-arm Navigation: a State of the Art Technology Comparison for Pedicle Screw Insertion
Brief Title: Mazor X Stealth Versus O-arm Navigation for Pedicle Screw Insertion
Acronym: RGNV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: P. D. Dr. med. Duccio BOSCHERINI (Other)
Responsible Party: Sponsor-Investigator, P. D. Dr. med. Duccio BOSCHERINI, Director of the Neuro Orthopedic Center, Neuro Orthopedic Center
Organization: Neuro Orthopedic Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-00305
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Disorder of Spine
Keywords: Vertebral instability; Spondylolisthesis; Discopathy
MeSH Terms: conditions — Spinal Diseases; Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: Medical device compared with gold standard
Who Masked: Participant
Masking Description: single-blind, only for the patient, after randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic group (RG) (Experimental): Patients in the RG group will be operated using the assistance of the Mazor X Stealth robot
  Interventions: Device: Guidance for pedicle screw insertion (Mazor Stealth)
- O-arm navigation group (NV) (Active Comparator): Patients in the NV group will be operated using the guidance of the Stealth navigation
  Interventions: Device: Guidance for pedicle screw insertion (O-arm Navigation)

INTERVENTIONS:
Device: Guidance for pedicle screw insertion (Mazor Stealth) — Using imaging devices and navigation for guidance, we perform a posterior vertebral fusion with pedicle screw insertion
  Arms: Robotic group (RG)
Device: Guidance for pedicle screw insertion (O-arm Navigation) — Using imaging devices and navigation for guidance, we perform a posterior vertebral fusion with pedicle screw insertion
  Arms: O-arm navigation group (NV)

SUMMARY:
The investigators would like to investigate the fluoro-registered Mazor X Stealth in terms of pedicle screw accuracy and radiation exposure in comparison with the O-arm and navigation as the institutional gold standard.

DETAILED DESCRIPTION:
Pedicle screw insertion for spinal fusion is a surgical procedure regularly performed around the world. Surgeons use free-hand, navigation or robotic techniques. The navigation began in 1995 in spine surgery. Surgical navigation systems provide pedicle screw insertion by projecting screw trajectories on a three-dimensional (3D) image acquisition, preoperatively or during the surgical procedure. Laine et al reported better accuracy and safety in pedicle screw insertion using the navigation system. Other authors reported less irradiation with the use of computer-assisted navigation. Robotic guidance was introduced in 2006 and assists the surgeon through a mechanical guidance according to a planning of screw trajectories on 3D imaging. This technique allows stable guidance for pedicle drilling and screw insertion, leading to greater screw positioning in lumbar fusion.

Medtronic (Medtronic, Minneapolis, MN, USA) introduced the Mazor X Stealth in Europa in 2019, including the Mazor robotic device with the navigation technology within the same system. The hypothesis would be a combination of the stability of the robot during screw insertion and the accuracy of the navigation with cumulative benefit from the two techniques.

The goal of this study is to compare radiological and clinical results of the use of the new Mazor Stealth with the surgical O-arm navigation during pedicle screw insertion for posterior lumbar fusion.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* who require pedicle screw insertion for vertebral posterior stabilization

Exclusion Criteria:

* children
* participants incapable of judgment
* participants under tutelage
* vertebral fusion indication without pedicle screw implantation
* refusal to participate
* data missing for radiation exposure calculation
* unstable vertebral fracture requiring urgent fixation
* pregnancy
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pedicle screw accuracy | Intraoperative
  Usinge the Heary classification for thoracic screws and the Gertzbein classification for lumbar screws

SECONDARY OUTCOMES:
Radiation exposure | Intraoperative
  Effective dose calculated with the PCXMC software for 2D (from dose area product) and with the ICRP 103 recommandations for 3D (from dose length product)

CONTACTS AND LOCATIONS:
Overall Officials: Duccio Boscherini, MD, PhD, Principal Investigator — Neuro Orthopedic Center
Locations (1):
- Neuro Orthopedic Center, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All data will be available for the Investigators and for control from the ethical commission if asked
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from the beginning of the study, and until 10 years according to cantonal rules
Access Criteria: Local professional computer
URL: https://www.cno.ch

REFERENCES:
- [Background] Staartjes VE, Molliqaj G, van Kampen PM, Eversdijk HAJ, Amelot A, Bettag C, Wolfs JFC, Urbanski S, Hedayat F, Schneekloth CG, Abu Saris M, Lefranc M, Peltier J, Boscherini D, Fiss I, Schatlo B, Rohde V, Ryang YM, Krieg SM, Meyer B, Kogl N, Girod PP, Thome C, Twisk JWR, Tessitore E, Schroder ML. The European Robotic Spinal Instrumentation (EUROSPIN) study: protocol for a multicentre prospective observational study of pedicle screw revision surgery after robot-guided, navigated and freehand thoracolumbar spinal fusion. BMJ Open. 2019 Sep 8;9(9):e030389. doi: 10.1136/bmjopen-2019-030389. PMID 31501123
- [Background] Nolte LP, Zamorano L, Visarius H, Berlemann U, Langlotz F, Arm E, Schwarzenbach O. Clinical evaluation of a system for precision enhancement in spine surgery. Clin Biomech (Bristol). 1995 Sep;10(6):293-303. doi: 10.1016/0268-0033(95)00004-5. PMID 11415570
- [Background] Staartjes VE, Klukowska AM, Schroder ML. Pedicle Screw Revision in Robot-Guided, Navigated, and Freehand Thoracolumbar Instrumentation: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Aug;116:433-443.e8. doi: 10.1016/j.wneu.2018.05.159. Epub 2018 May 31. PMID 29859354
- [Background] Laine T, Lund T, Ylikoski M, Lohikoski J, Schlenzka D. Accuracy of pedicle screw insertion with and without computer assistance: a randomised controlled clinical study in 100 consecutive patients. Eur Spine J. 2000 Jun;9(3):235-40. doi: 10.1007/s005860000146. PMID 10905443
- [Background] Hartl R, Lam KS, Wang J, Korge A, Kandziora F, Audige L. Worldwide survey on the use of navigation in spine surgery. World Neurosurg. 2013 Jan;79(1):162-72. doi: 10.1016/j.wneu.2012.03.011. Epub 2012 Mar 30. PMID 22469525
- [Background] Lieberman IH, Togawa D, Kayanja MM, Reinhardt MK, Friedlander A, Knoller N, Benzel EC. Bone-mounted miniature robotic guidance for pedicle screw and translaminar facet screw placement: Part I--Technical development and a test case result. Neurosurgery. 2006 Sep;59(3):641-50; discussion 641-50. doi: 10.1227/01.NEU.0000229055.00829.5B. PMID 16955046
- [Background] Togawa D, Kayanja MM, Reinhardt MK, Shoham M, Balter A, Friedlander A, Knoller N, Benzel EC, Lieberman IH. Bone-mounted miniature robotic guidance for pedicle screw and translaminar facet screw placement: part 2--Evaluation of system accuracy. Neurosurgery. 2007 Feb;60(2 Suppl 1):ONS129-39; discussion ONS139. doi: 10.1227/01.NEU.0000249257.16912.AA. PMID 17297375
- [Background] Schroder ML, Staartjes VE. Revisions for screw malposition and clinical outcomes after robot-guided lumbar fusion for spondylolisthesis. Neurosurg Focus. 2017 May;42(5):E12. doi: 10.3171/2017.3.FOCUS16534. PMID 28463610
- [Background] Heary RF, Bono CM, Black M. Thoracic pedicle screws: postoperative computerized tomography scanning assessment. J Neurosurg. 2004 Apr;100(4 Suppl Spine):325-31. doi: 10.3171/spi.2004.100.4.0325. PMID 15070139
- [Background] Gertzbein SD, Robbins SE. Accuracy of pedicular screw placement in vivo. Spine (Phila Pa 1976). 1990 Jan;15(1):11-4. doi: 10.1097/00007632-199001000-00004. PMID 2326693
- [Background] The 2007 Recommendations of the International Commission on Radiological Protection. ICRP publication 103. Ann ICRP. 2007;37(2-4):1-332. doi: 10.1016/j.icrp.2007.10.003. PMID 18082557
- [Background] Servomaa A, Tapiovaara M. Organ dose calculation in medical x ray examinations by the program PCXMC. Radiation protection dosimetry. 1998 Nov 1;80(1-3):213-9
- [Background] Nuclear Energy Agency Forum on Stakeholder ConfidenceChilton Seminar: Roger Cox -'Risks from low doses of low-LET radiation - the US National Academy of Sciences BEIR VII report'SRP Meeting on Source ManagementScientific Symposium to Mark the Past and Future Achievements of Richard Doll. Journal of Radiological Protection. 2006;26(1):119-123
- See also: [Internet]. Medtronic.com. 2019 [cited 15 January 2020]. — https://www.medtronic.com/us-en/healthcare-professionals/products/neurological/spine-robotics/mazorx.html